CLINICAL TRIAL: NCT00050765
Title: A Phase I Multi-Center Study to Assess the Safety and Cardiovascular Effects of MyoCell™ Implantation in Patients With a Previous MI and Placement of an ICD Requiring De Novo Coronary Artery Bypass Graft Therapy
Brief Title: Autologous Cultured Myoblasts (BioWhittaker) Transplanted Via Myocardial Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bioheart, Inc. (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Protocol BMI-US-01-001; Version F
Record Dates: First submitted 2002-12-18; First posted 2002-12-19 (Estimated); Last update posted 2006-03-08 (Estimated); Status verified 2006-03

CONDITIONS: Congestive Heart Failure; Coronary Artery Disease; Myocardial Infarction
Keywords: Myocardial Infarction; Heart disease; Coronary bypass graft (CABG) surgery; Implantable Cardioverter Defibrillator (ICD); CABG; ICD; Heart failure
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease; Myocardial Infarction; Heart Diseases

INTERVENTIONS:
Drug: MyoCell™ Autologous Myoblasts

SUMMARY:
MyoCell™ implantation by epicardial injection during CABG surgery has the potential to add a new dimension to the management of post-infarct deterioration of cardiac function. Based on existing non-clinical studies and clinical reports, implantation of autologous skeletal myoblasts appears to lead to the replacement of non-functioning myocardial scar with functioning muscle and appears to improve myocardial performance relative to case without myoblast implantation. In a few investigational patients, myoblast implantation can be, and has been, done in conjunction with CABG and appears to have the potential to provide for additive treatment during surgery. The present study is being conducted to evaluate more fully the safety of MyoCell™ implantation via epicardial injection during CABG surgery and its effect on regional myocardial function.

DETAILED DESCRIPTION:
MyoCell™ mediated cellular cardiomyoplasty is a novel therapeutic approach to the management of progressive heart failure in patients who have damaged myocardial tissue resulting from a myocardial infarct. MyoCell™ consists of patient autologous skeletal myoblasts which are expanded ex vivo and supplied as a cell suspension in a buffered salts solution for injection into the area of damaged, akinetic myocardium with the goal of having the myoblasts populate the implant area and generate elastic, contractile skeletal muscle-like tissue within the damaged myocardium. Because the physiological goal is to replace inelastic, fibrous myocardial scar tissue with skeletal muscle-like tissue, originating from the cellular implants, this therapeutic approach is termed "cellular cardiomyoplasty" or "CCM".

The purpose of this trial is to assess the safety of MyoCell™(expanded autologous skeletal myoblasts) using a dose escalation methodology following epicardial injection into myocardial scar tissue in patients who have experienced anterior, lateral, posterior or inferior wall myocardial infarction, require coronary artery bypass graft (CABG) surgery and who have an implantable cardioverter defibrillator (ICD) in place (ICD can be implanted during the CABG procedure or 3 to 4 days post CABG procedure). Safety endpoints will be the evaluation of the nature and frequency of Adverse Events during the 12-month period following MyoCell™ treatment.

If a patient meets the baseline enrollment criteria, a 5-10 gram skeletal muscle biopsy will be obtained for myoblast isolation and expansion in vitro at Bioheart's designated facility for MyoCell™ production. Biopsy will occur 3 - 4 weeks prior to the anticipated implantation of the MyoCell™ product. At the time of the patient's CABG surgery MyoCell™ will be injected into the akinetic myocardial scar in the region of a previous infarct utilizing a sterile hypodermic syringe fitted with a 25 gauge needle.

This will be a dose escalation study with 3 cohort groups consisting of 5 patients each. A report of the 1 month safety data from each cohort will be presented to the data safety monitoring board for permission to go to the next higher dosage. In the first cohort of this dose escalation study; 2 injections will be performed, for the second cohort; 6 injections and for the third cohort; 18 injections depending on the size of the infarct scar, so as to inject the entire myocardial infarct scar akinetic area.

ELIGIBILITY:
Inclusion Criteria:

* Defined region of myocardial dysfunction related to previous myocardial infarction involving the anterior, lateral, posterior or inferior walls, > 12 weeks old at the scheduled time of MyoCell™ implantation procedure
* Patients must have an implantable cardioverter defibrillator (ICD) in place or, patients must receive ICD placement during the CABG procedure or 3 to 4 days after the CABG procedure
* Planned CABG procedure for revascularization
* Heart failure patient in New York Heart Association Symptom Class 2 or 3 who is on optimal medical therapy
* Age > 18 and < 80 years
* Able to undergo surgical biopsy of the skeletal muscle and successful culture of the harvested myoblasts
* Target region wall thickness > 6 mm by echocardiography
* Left ventricular ejection fraction > 20% and < 40% by radionuclide ventriculography or left ventricular angiography at screening
* If a female of childbearing potential, urine pregnancy test must be negative
* Able to give written informed consent

Exclusion Criteria:

* Patient medically unable to undergo CABG surgery
* Any patient who has had a documented myocardial infarction (ECG changes or elevated cardiac enzymes consistent with MI) within 30 days of the scheduled surgical revascularization and cellular implantation procedure.
* Known sensitivity to gentamicin sulfate and/or amphotericin-B
* Exposure to any investigational drug or procedure within 4 weeks prior to study entry
* The use or expected use of antineoplastic drugs
* History of skeletal muscle disease, either primary (i.e., myopathy) or secondary (i.e., ischemic) or any underlying myopathy such as myasthenia gravis, muscular dystrophy, etc.) as determined by a board certified pathologist examining sample of patients muscle biopsy
* Previous angiogenic therapy and/or myocardial laser therapy
* History of cancer within 5 years, except for basal cell carcinoma of the skin
* PSA suggestive of carcinoma of the prostate (i.e., > 4)
* Patient with CEA >2.5 ng/mL or end stage renal disease
* Patients with active infectious disease and/or who are known to have tested positive for HIV, HTLV, HBV-sAg, HCV, CMV and/or syphilis. If the panel includes antibodies to the HBc and HBV-sAg, then an expert will be consulted.
* Females who are pregnant or nursing. Females of childbearing potential must be using to the investigator's satisfaction, a medically accepted method of birth control (e.g., but not limited to, oral or implanted contraceptive therapy or intrauterine devices) and agree to continue for the duration of the study.
* Any illness which might affect patient's survival over the study follow-up period
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results.
* Patient with an any previous cardiac surgery
* Patient with valvular disease greater than mild in degree which is considered the primary cause of their heart failure
* Patient in New York Heart Association Symptom Class 1 or 4
* Patient with serum creatinine > 2.5
* No informed consent or unable to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2006-08; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Bioheart, Inc, Fort Lauderdale, Florida
  - ACRI, Atlanta, Georgia
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Mt. Sinai Medical Center, New York, New York
  - Duke University, Durham, North Carolina

REFERENCES:
- See also: Bioheart Inc. website — http://bioheartinc.com